CLINICAL TRIAL: NCT01872858
Title: Efficacy and Safety of Cilostazol in Patients of Vascular Cognitive Impairment-no Dementia (VCIND)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Jianhui Fu, Department of Neurology, Huashan Hospital, Huashan Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: jianhuifu2013; NCT01862575 (obsolete NCT alias)
Record Dates: First submitted 2013-06-05; First posted 2013-06-07 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Aspirin; Cilostazol

ARMS (2):
- Aspirin (Active Comparator): Aspirin, 100mg, Q.D, p.o, 2yr
  Interventions: Drug: Aspirin
- Cilostazol (Experimental): cilostazol, 100mg, B.I.D, p.o, 2yr
  Interventions: Drug: Cilostazol

INTERVENTIONS:
Drug: Aspirin — Aspirin, 100mg, Q.D, p.o, 2yr
  Arms: Aspirin
Drug: Cilostazol — cilostazol, 100mg, B.I.D, p.o, 2yr
  Arms: Cilostazol

SUMMARY:
Patients of vascular cognitive impairment-no dementia (VCIND) in one group is prescribed cilostazol,in the other group is prescribed aspirin. Evaluate both of them in cognitive function, MRI and other sides at given time. The investigators hypothesize that cilostazol is more efficient and safer than aspirin in patients with VCIND.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 50-80, both gender；
2. Small vessel disease and associated cognitive impairment, diagnosed as VCIND；
3. Non-specific subjective symptoms (dizziness, somnolence, numbness in limbs) are acceptable.
4. Normal hepatic and renal function.
5. With good compliance.

Exclusion Criteria:

1. Aged above 80 or less than 50.
2. Dementia.
3. Cerebral infarction(>2cm).
4. Major vascular lesion. (stenosis>50%).
5. Cardiac cerebral infarction.
6. Intracerebral Hemorrhage.
7. Clinical manifestations cannot attribute to small vessel disease.
8. Major depression or dysfunction in speech, visual ability, hearing or aphasia that would interfere with the cognitive assessment.
9. Severe systematic organic impairment(cardiac, hepatic, renal dysfunction).
10. Thrombocytopenic Purpura.
11. History of hemorrhage in digestive system or surgery in past 3 months.
12. Previously on cilostazol treatment for more than 3 month.
13. Allergic to aspirin or cilostazol.
14. Enrolled in other clinical trials in past 3 months.
15. Lack of informed consent or compliance.
16. Contraindications for MRI scan.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-11; Primary Completion 2012-11 (Actual); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
changes in cognitive function | baseline, 3month, 6month, 1year, and 2year
  scores in Montreal Cognitive Assessment，Mini-Mental Status Examination, Clinal Dementia Rating，trail making test, similarity test, Stroop test.

SECONDARY OUTCOMES:
Number of Participants with Incident cerebral vascular event | 3month, 6month, 1year and 2year
  including cerebral infarct, cerebral hemorrhage, transient ischemic attack.
Changes of peripheral inflammatory markers level | baseline, 2year
  intercellular adhesion molecules(ICAM), thrombomodulin, tissue factor(TF), tissue factor plasma inhibitor，TFPI, etc.
The progression of cerebral white matter lesion and lacunar infarction | baseline, 3month, 6month, 1year and 2year
changes in MRI-diffused tension image(DTI) | baseline, 2year
  cerebral volume , lacune infarct, white matter lesion, micro-bleed, apparent diffusion coefficient(ADC) .

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Neurology, Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China